CLINICAL TRIAL: NCT05175495
Title: To Study the Risk Factors of Youth Coronary Heart Disease From Inflammatory Cytokines，Lifestyle and Familial Inheritance
Brief Title: Influencing Factors of Coronary Heart Disease in Young People
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hongzhuan Sheng (Other)
Collaborators: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor-Investigator, Hongzhuan Sheng, Chief physician, Affiliated Hospital of Nantong University
Organization: Affiliated Hospital of Nantong University (Other)
Other Study IDs: Observational
Record Dates: First submitted 2021-11-05; First posted 2022-01-03 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Coronary Heart Disease
Keywords: Coronary heart disease; Inflammatory cytokines; lifestyle; Familial inheritance; Myocardial infarction
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood、serum、plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal young: Aged less than 45 years old,no underlying heart disease
- Young people diagnosed with coronary heart disease: Aged less than 45 years old,Diagnosed coronary heart disease;Confirmed by coronary angiography;Diagnosed myocardial infarction;Typical symptom of ischemic chest pain with positive stress test;
- Coronary heart disease: Older than 65 years, diagnosed with coronary heart disease

SUMMARY:
The incidence of coronary heart disease in young people is not uncommon and the investigators will explore the factors contributing to this outcome

DETAILED DESCRIPTION:
Through the multi-center clinical research conducted by several units in Nantong city, the risk factors and aggregation of the incidence of CHD among young people in nantong city were obtained, so as to fill in the blank of domestic multi-center research and reduce the incidence of CHD among young people.The investigators will conduct a long-term follow-up study on the young patients with CHD to screen the factors contributing to the poor prognosis of CHD in young patients.The investigators will fill this gap and intervene early to improve patients' quality of life and prolong their survival

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed coronary heart disease
* Confirmed by coronary angiography
* Diagnosed myocardial infarction
* Willing to sign an inform consent

Exclusion Criteria:

* Patients won't sign an inform consent or will not comply with the follow up.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Diagnosed coronary heart disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Whether inflammatory factors are differentially expressed in young patients with coronary heart disease | Until April 2024
  The Investigators will analyze blood samples from the participants to see if there was a difference in the expression of inflammatory factors with high correlation compared with the control group by ELESA and High-throughput sequencing.
The effect of gene activity on youth morbidity | Until April 2024
  The investigators will use enrichment analysis to screen the target genes and sequence the participants.Whether the target gene was expressed at high levels in the participants.And the investigators will further analyze the target gene
Sedentary, high-fat diet, lack of exercise and other unhealthy lifestyle effects on young people | Until April 2024
  The researchers will retrospectively examine the participants' negative lifestyle habits, such as sedentary behavior, smoking, high-fat diet, and lack of exercise, in combination with their coronary angiography results

CONTACTS AND LOCATIONS:
Overall Officials: hzh sheng, Dr., Study Chair — Affiliated Hospital of Nantong University
Locations (1):
- shengHz, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
We will share our findings with you when the 2024 project is due